CLINICAL TRIAL: NCT05667272
Title: A Study on the Occurrence Time of Clinically Relevant Postoperative Pancreatic Fistula of Grade-B After Pancreatoduodenectomy
Brief Title: A Study on the Occurrence Time of Grade-B Pancreatic Fistula After Pancreatoduodenectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changzhou Second People's Hospital affiliated with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SYuhang
Record Dates: First submitted 2022-12-19; First posted 2022-12-28 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Postoperative Pancreatic Fistula
Keywords: postoperative pancreatic fistula

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pancreatic fistula group: no intervention(s)
  Interventions: Other: No intervention
- non-pancreatic fistula group: no intervention(s)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
To confirm the time point of CR-POPF of grade-B that patients with biochemical leak after PD or LPD turned into.

DETAILED DESCRIPTION:
1. To confirm the time point of CR-POPF of grade-B that patients with biochemical leak after PD or LPD turned into.
2. Establishment of risk assessment model for Grade B fistula.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent Pancreatoduodenectomy (PD) or Laparoscopic pancreatoduodenectomy (LPD) surgery.
* Surgery performed by the same surgical team.

Exclusion Criteria:

* PD or LPD combined with another organ resection.
* PD or LPD performed due to trauma.
* PD or LPD for emergency treatment, such as the rupture and bleeding of tumor.
* Palliative resection.
* Patients with severe organ dysfunction before surgery.
* Patients treated with preoperative neoadjuvant chemotherapy or other treatments (Radiotherapy, targeted immunotherapy, etc.).
* Patients with missing data for clinical or radiographic variables.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: (1) Patients with PD or LPD surgery; (2) Surgery performed by the same surgical team.
Sampling Method: Non-Probability Sample
Enrollment: 216 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | up to postoperative 30 days
  Postoperative complications for each patient

CONTACTS AND LOCATIONS:
Overall Officials: chunfu zhu, PhD, Study Chair — Changzhou Second People's Hospital
Locations (1):
- Changzhou Second People's Hospital affiliated to Nanjing Medical University, Changzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bassi C, Marchegiani G, Dervenis C, Sarr M, Abu Hilal M, Adham M, Allen P, Andersson R, Asbun HJ, Besselink MG, Conlon K, Del Chiaro M, Falconi M, Fernandez-Cruz L, Fernandez-Del Castillo C, Fingerhut A, Friess H, Gouma DJ, Hackert T, Izbicki J, Lillemoe KD, Neoptolemos JP, Olah A, Schulick R, Shrikhande SV, Takada T, Takaori K, Traverso W, Vollmer CM, Wolfgang CL, Yeo CJ, Salvia R, Buchler M; International Study Group on Pancreatic Surgery (ISGPS). The 2016 update of the International Study Group (ISGPS) definition and grading of postoperative pancreatic fistula: 11 Years After. Surgery. 2017 Mar;161(3):584-591. doi: 10.1016/j.surg.2016.11.014. Epub 2016 Dec 28. PMID 28040257